CLINICAL TRIAL: NCT03048643
Title: CATS-CARE: Combining Opioid Addiction Treatment Services With CARe for Infectious Endocarditis
Brief Title: Combining Opioid Addiction Treatment Services With CARe for Infectious Endocarditis
Acronym: CATS-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Fanucchi (Other)
Responsible Party: Sponsor-Investigator, Laura Fanucchi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-1001-F1V
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Endocarditis, Bacterial; Opioid-use Disorder; Buprenorphine; Outpatient Parenteral Antibiotic Therapy
MeSH Terms: conditions — Endocarditis, Bacterial; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Subjects will receive medication-assisted treatment for opioid use disorder and will complete IV antibiotic therapy for infective endocarditis according to usual care.
- Outpatient Parenteral Antibiotic Therapy (Experimental): Subjects will receive medication-assisted treatment for opioid use disorder and will complete IV antibiotic therapy via outpatient parenteral antibiotic therapy (OPAT).
  Interventions: Behavioral: Outpatient parenteral antibiotic therapy

INTERVENTIONS:
Behavioral: Outpatient parenteral antibiotic therapy — Subjects randomized to OPAT will complete IV antibiotic therapy for infective endocarditis as an outpatient according to published guidelines.
  Other Names: OPAT
  Arms: Outpatient Parenteral Antibiotic Therapy

SUMMARY:
Hospitalizations for severe infections associated with opioid use disorder (OUD), such as infective endocarditis (IE), have doubled in the US over the past decade and are frequently prolonged and resource-intensive. Once medically stabilized, persons with IE but without drug use typically enroll in outpatient parenteral antibiotic therapy (OPAT), while persons with IE and OUD are kept in the hospital for the duration of therapy (often 6 weeks or more) largely due to concerns of ongoing drug use. Unfortunately, hospitalization for IE with OUD infrequently includes evidence-based medication-assisted treatment (MAT) with buprenorphine or methadone to address the OUD, despite the strong evidence that MAT decreases illicit drug use and mortality. Enrolling hospitalized persons with IE due to OUD into comprehensive MAT (i.e., buprenorphine + counseling) while inpatient, and providing an intensive transitional outpatient care program supporting MAT, may support provision of outpatient IV antibiotic therapy and be cost effective. The primary aim of this pilot randomized clinical trial is to evaluate the equivalence of current practice plus buprenorphine (keeping patients with IE due to opioid use disorder in the hospital for the full duration of antibiotic treatment) compared to OPAT plus buprenorphine (discharge with outpatient treatment once medically stable).

ELIGIBILITY:
Inclusion Criteria:

* meeting OUD by DSM-V criteria
* have IE by Duke's criteria
* candidates for outpatient treatment with buprenorphine
* accepting of buprenorphine treatment
* anticipated to be discharged home after medically stabilized
* requiring ≥ 2 weeks of IV antibiotic therapy
* having ≥ 1 week of IV antibiotic therapy remaining at the time of medical readiness for discharge (as defined by the primary clinical team),
* and providing informed consent.

Exclusion Criteria:

* presence of stroke or central nervous system involvement
* clinically active embolic sequelae (e.g. pulmonary sepsis, mycotic aneurysms, splenic abscesses)
* TV treated surgically or endovascularly (AngioVac)
* presence of osteomyelitis
* fungal IE
* patients who require inpatient physical rehabilitation determined by physical or occupational therapy assessment
* current pregnancy
* current severe methamphetamine, cocaine, alcohol or benzodiazepine use disorders by DSM-V criteria
* currently enrolled in ongoing MAT for OUD
* hypersensitivity or allergy to buprenorphine
* chronic pain requiring opioids
* class III or IV heart failure
* cirrhosis
* end stage renal disease
* other significant screening laboratory/medical/psychiatric/psychosocial condition that may prevent the volunteer from safely participating in the study in the opinion of the investigator (e.g. currently suicidal)
* pending legal action that could interfere with study participation
* living more than a 45-minute drive from UK given the intense outpatient component to the intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Illicit drug use | 12 weeks after discharge
  Participants will be asked by their clinician to self report illicit drug use at their follow up visit 12 weeks after discharge

SECONDARY OUTCOMES:
Completion of recommended IV antibiotic therapy | 12 weeks after discharge
  Participants will be asked by their clinician to self report compliance to the recommended IV antibiotic therapy at their follow up visit 12 weeks after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Laura Fanucchi, MD, Principal Investigator — University of Kentucky; Sharon Walsh, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanucchi LC, Walsh SL, Thornton AC, Nuzzo PA, Lofwall MR. Outpatient Parenteral Antimicrobial Therapy Plus Buprenorphine for Opioid Use Disorder and Severe Injection-related Infections. Clin Infect Dis. 2020 Mar 3;70(6):1226-1229. doi: 10.1093/cid/ciz654. PMID 31342057